CLINICAL TRIAL: NCT04529265
Title: Effectiveness and Safety of Methylene Blue for Prevention of Postoperative Neurocognitive Disorders in Patients Undergoing Pancreatic Tumor Surgery: A Prospective Randomized Controlled Clinical Trial
Brief Title: Methylene Blue and Postoperative Neurocognitive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2008222-Exps
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylene Blue group (Experimental): The first dosage: 2mg/kg MB diluted with normal saline into total 50 ml volume intravenous administration after induction of anesthesia within one hour; The second dosage: 1mg/kg MB diluted with normal saline into total 50 ml volume intravenous administration before the end of surgery within 30 minutes.
  Interventions: Drug: Methylene Blue
- Control group (Placebo Comparator): The first dosage: normal saline in total 50 ml volume intravenous administration after induction of anesthesia within one hour; The second dosage: normal saline in total 50 ml volume intravenous administration before the end of surgery within 30 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylene Blue — Intraoperative infusion of 2mg/kg MB after induction of anesthesia for 1 h and 1mg/kg MB with 30 min before the end of surgery
  Arms: Methylene Blue group
Drug: Placebo — Equal volume of normal saline after induction of anesthesia for 1 h and Equal volume of normal saline within 30 min before the end of surgery
  Arms: Control group

SUMMARY:
Postoperative Neurocognitive Disorders are the most common neurological complications after major surgery, which are associated with higher increased mortality and morbidity in elderly patients undergoing major surgery. Until now highly effective intervention has not been established yet. Recent preclinical studies suggest neuroinflammation may be linked to pathogensis of (postoperative delirium) POD and postoperative cognitive dysfunction (POCD). As Methylene blue(MB) has neuroprotective and anti-inflammatory properties, and it is a safe drug with long history of clinical use, we propose that inflammation-targeted interventions may be useful to prevent POD/POCD in surgical patients.

DETAILED DESCRIPTION:
Pancreatic cancer is one of the most common incident cancers that causes cancer death in China. The patients undergoing pancreatic cancer surgery not only have a low survival rate, but also have high postoperative complications, including postoperative delirium(POD) characterized by an acute change in cognition with altered consciousness and impaired attention, and postoperative cognitive dysfunction(POCD) mainly manifested as reduced ability of learning and memory. It is reported that POD occurred in 10% - 60% of elderly surgical patients, varying by surgical procedure, while the incidence of POCD is approximately 25%-40%. Although it was reported that small dosage of intravenous dexmedetomidine maybe reduce the incidence of POD/POCD, a large number of studies had also shown that dexmedetomidine would promote breast cancer, liver cancer and lung cancer cells' proliferation and migration, which urged to find more effective and safer treatment strategies to reduce the incidence of postoperative neurocognitive dysfunction in elderly cancer patients.

The preclinical and clinical studies have demonstrated anesthesia/surgery-induced neuroinflammation and oxidative stress are strongly associated with postoperative neurocognitive disorders. The systemic inflammation plays a central role in neurodegenerative diseases, leading to neuronal death, metabolic disturbance, and excessive reactive oxidative species(ROS) production. Actually, recent experimental evidences have linked anesthesia/surgery-induced inflammation to POCD, and the available data support that restoration of neuroinflammation could reduce postoperative cognitive impairments in developing and aging animals. Therefore, we propose those inflammation-targeted interventions may be useful to prevent POD/POCD in elderly surgical patients.

Methylene blue(MB) is a diaminophenothiazine with a long history of clinical use due to its safe profile. The studies have indicated that MB, as a redox mediator in the electron transfer chain (ETC), restores mitochondrial function and enhances brain metabolism. In recent years its role as a mitochondrial protective agent has elicited much of its renewed interest, especially its neuroprotective effects in clinical studies against ischemic stroke, chemotherapy-induced encephalopathy and neurodegenerative disorders associated with psychoses. MB has been proposed to protect selective regions of the brain, wherein memory is encoded and processed in various models of brain dysfunction-induced amnesia, and importantly, enhances learning and memory in patients with mental diseases and healthy human through its beneficial brain network effects. Now its emerging role as neuroprotection and memory-enhancer makes this old drug become a promising cure for neurodegenerative diseases. Our previous clinical study ( NCT04341844) found that the single dosage of 2mg/kg MB was safe to the elderly patients undergoing non-cardiac surgery, and was effective to prevent of the incidence of POD and early POCD. And our experimental study also found that MB inhibited neuroinflammation and improved neurobehavioral deficits in lipopolysaccharide-treated mice via inhibiting the microglial Siah2/Morg1/PHD3 pathway. However, whether the safety and effectiveness of MB could prevent postoperative cognitive impairments in pancreatic tumor patients needs further investigation. Therefore, we design this prospective randomized controlled clinical trial to test whether MB could decrease the incidence of POD/POCD in patients undergoing pancreatic tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged 55-80 years old
* planning to undergo pancreatic tumor surgery.
* Patients have the ability to act in full spirit, understand and sign the informed consent, and are willing to complete the whole research process.

Exclusion Criteria:

* preexisted dementia, major depression or other serious mental or neurological disorders
* history of allergy to MB or 6-phospho-glucose dehydrogenase deficiency (favism)
* MMSE<24
* illiterate patients
* patients diagnosed with rheumatoid diseases such as systemic lupus erythematosus, rheumatoid arthritis and ankylosing spondylitis
* drug or alcohol abuse or recent drug administration that may lead to drug interactions, such as selective serotonin reuptake inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitors (SNRIs)
* history of major head trauma
* serious medical diseases (ie. heart failure, pulmonary hypertension, acute stage of myocardial infarction or respiratory failure, hepatic and renal dysfunctions)
* severe language, visual or auditory deficiency
* other neoplastic diseases diagnosed in the past 5 years
* participated in other clinical trials within 3 months.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium(POD) | Participants will be followed for the duration of hospital stay, an expected average of 7 days.
  the effectiveness of MB in reducing the incidence of POD compared with placebo in patients undergoing pancreatic tumor surgery.

SECONDARY OUTCOMES:
type and duration of POD | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Safety Assessments: incidence of perioperative adverse events | the whole perioperative period
  the incidence of perioperative adverse events to reflect safety of MB administration
neuroinflammation biomarkers | on the day of surgery (before anesthesia and at the end of surgery) and postoperative one day
  the changes in levels of neuroinflammation biomarkers ( IL-6 and IL-8 )between MB group and control group
expressions of inflammatory and adhesion genes in cerebral endothelial cells | before anesthesia and at first day after surgery
  TNF-α, monocyte chemoattractant protein-1 (MCP-1), Claudin 5 (CLND5) and adhesion factors including vascular cell adhesion protein 1 (VCAM-1) and intercellular adhesion molecule 1 (ICAM-1)
numbers of PBMCs adhesion to cerebral endothelial cells | before anesthesia and at first day after surgery
Incidence of postoperative cognitive dysfunction (POCD) | Up to the 7th day after surgery
  the effectiveness of MB in reducing the incidence of POCD compared with placebo in patients undergoing pancreatic tumor surgery.
overall survival | up to 3 years after surgery
  the effectiveness of MB on overall survival compared with placebo in patients undergoing pancreatic tumor surgery.
disease-free survival | up to 3 years after surgery
  the effectiveness of MB on disease-free survival compared with placebo in patients undergoing pancreatic tumor surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deng Y, Wang R, Li S, Zhu X, Wang T, Wu J, Zhang J. Methylene blue reduces incidence of early postoperative cognitive disorders in elderly patients undergoing major non-cardiac surgery: An open-label randomized controlled clinical trial. J Clin Anesth. 2021 Feb;68:110108. doi: 10.1016/j.jclinane.2020.110108. Epub 2020 Oct 19. PMID 33091706
- [Background] Deiner S, Luo X, Lin HM, Sessler DI, Saager L, Sieber FE, Lee HB, Sano M; and the Dexlirium Writing Group; Jankowski C, Bergese SD, Candiotti K, Flaherty JH, Arora H, Shander A, Rock P. Intraoperative Infusion of Dexmedetomidine for Prevention of Postoperative Delirium and Cognitive Dysfunction in Elderly Patients Undergoing Major Elective Noncardiac Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 Aug 16;152(8):e171505. doi: 10.1001/jamasurg.2017.1505. Epub 2017 Aug 16. PMID 28593326
- [Background] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Background] Tucker D, Lu Y, Zhang Q. From Mitochondrial Function to Neuroprotection-an Emerging Role for Methylene Blue. Mol Neurobiol. 2018 Jun;55(6):5137-5153. doi: 10.1007/s12035-017-0712-2. Epub 2017 Aug 24. PMID 28840449
- [Background] Gonzalez-Lima F, Barksdale BR, Rojas JC. Mitochondrial respiration as a target for neuroprotection and cognitive enhancement. Biochem Pharmacol. 2014 Apr 15;88(4):584-93. doi: 10.1016/j.bcp.2013.11.010. Epub 2013 Dec 4. PMID 24316434
- [Background] Wischik CM, Staff RT, Wischik DJ, Bentham P, Murray AD, Storey JM, Kook KA, Harrington CR. Tau aggregation inhibitor therapy: an exploratory phase 2 study in mild or moderate Alzheimer's disease. J Alzheimers Dis. 2015;44(2):705-20. doi: 10.3233/JAD-142874. PMID 25550228